CLINICAL TRIAL: NCT04268810
Title: Prospective Randomised Trial Comparing Intravesical Chondroitin Sulphate 2% and DMSO in the Treatment of Painful Bladder Syndrome/ Interstitial Cystitis
Brief Title: Prospective Trial Comparing Intravesical Chondroitin Sulphate 2% and DMSO in the Treatment of PBS/Interstitial Cystitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: too many side effect in the control arm (DMSO)
Sponsor: National Multiple Sclerosis Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S52212; Uracyst study (Other: KU Leuven)
Record Dates: First submitted 2013-03-31; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Painful Bladder Syndrome; Interstitial Cystitis
Keywords: painful bladder syndrome; interstitial cystitis; chondroitin sulphate; DMSO
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Administration, Intravesical

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chondroitin sulphate 2% (Experimental): chondoritin sulphate 2% ( Uracyst) for bladder instillation. One bladeer instillation per week during 6 weeks.
  Interventions: Procedure: Bladder instillations
- DMSO 50% (Active Comparator): DMSO 50% in saline for bladder instillation. One bladder instillation per week during 6 weeks
  Interventions: Procedure: Bladder instillations

INTERVENTIONS:
Procedure: Bladder instillations — bladder instillations with either solution (DMSO or Uracyst)

SUMMARY:
Painful bladder syndrome/interstitial cystitis (PBS/IC)is a disease of unknown origin with a significant impact on the quality of life. Next to oral treatment with tricyclic antidepressants or pentosan polysulphate, intravesical treatment can be used as well. The purpose of this treatment is to restore the protective lining of the bladder that consists of glycan structures (GAG). Currently only dimethylsulfoxide (DMSO) is FDA approved for this. Several other compounds have been introduced. We want to compare a solution of chondroitin sulphate 2% with the standard DMSO solution. We will compare the patient perception of benefit,but also pain scores, quality of life and micturition diaries.

DETAILED DESCRIPTION:
A. Introduction

Painful bladder syndrome(PBS) is a syndrome which is poorly understood. Patients usually report suprapubic pain related to bladder filling and also report urinary urgency and frequency. In a subgroup of patients, typical cystoscopic findings can be noted and this defines this subgroup as interstitial cystitis. (Abrams et al. 116-26) The treatment of PBS/IC is empirical. Bladder hydrodistension under anesthesia, tricyclic antidepressants, antihistaminics and intravesical DMSO instillations are the only treatment for which some evidence exists in the literature. More than 150 other treatment modalities have been described . Most of them were poorly studied. (Fall et al. 1-99) Intravesical treatment with DMSO has stood the test of time and is the only FDA approved intravesical treatment of PBS/IC. DMSO however is also used as a solvent in the chemical industry and is in fact used ' off label' in this indication. (Erickson 333-43;Emerson and Perezmarrero A136;Perez-Marrero, Emerson, and Feltis 36-39) One of the theories on which intravesical treatment is based, claims that the glycosaminoglycan layer, which protects the urothelial cells is damaged. DMSO, Chondroitin sulphate, hyaluronic acid and heparin have been used to repair the GAG layer with variable clinical success. (Daha et al. 369-72;Daha et al. 987-90;Riedl et al. 717-21) Chondroitin sulphate seems to be promising, but comparative data are lacking. (Gauruder-Burmester and Popken 355-59;Nickel et al. 56-60;Hauser et al. 2477-82;Nordling and van Ophoven 328-35) Assessing the outcome of such treatments is difficult. Objective parameters such as daytime and nighttime frequency may not always reflect the impact of the condition on the life of the patient.

Patient reported outcome parameters are more frequently used to assess treatments in overactive bladder disease and in painful bladder research. Several validated questionnaires can be used to assess patients with PBS/IC. One of the most frequently used is the O'Leary-Sant questionnaire ( see annex 1). Next to this questionnaire the Global Response Assessment will be used. This is a validated 7 point Likert scale comparing the current status of the patient to the pre-intervention status. This scale has been used in several other studies on PBS/IC. (Nickel et al. 910-18;Baranowski et al. 33-36) Aim To compare the clinical effectiveness of intravesical chondroitin sulphate 2% ( Uracyst ™) and DMSO 50% in the treatment of patients with painful bladder syndrome

B. Randomization A central randomization will be used. Participating centers will have to contact the trial office of the dept. of urology of the University Hospitals Leuven to randomize the patient to one or the other treatment, either by telephone 016/346692 or 016/348345 or by mail elza.goossens@uzleuven.be or evelien.vankriekingen@uzleuven.be . A block randomization per center will be done. The randomization list was generated on a web application ( www.randomizer.org) to ensure an unbiased randomization schedule.

C. Protocol of administration Patients that are enrolled in the study will receive one intravesical instillation of Uracyst or DMSO a week during 6 weeks. DMSO is prepared as a 50% solution in 50cc physiologic serum. Uracyst will be prepared by the nurse or urologist administering the product.

Uracyst is delivered as a 2% sterile solution in 20cc vials. The instillation is done by a urethral catheterization. The catheter is withdrawn once the fluid has been instilled. The solution is kept in the bladder for at least 30 minutes. A simple instillation protocol is followed, meaning that the patient can move immediately after the instillation of the product. The product is eliminated by spontaneous voiding after 30 minutes.

D. Safety Safety is assessed by monitoring adverse events at every visit. Anticipated adverse events are hematuria, algiuria, urinary tract infection and garlic odor ( for DMSO)…

E. Statistics Comparison of the mean GRA by T-test will be used for the primary endpoint. Appropriate statistical tests will be used for the secondary variables.

To detect a 0.75 difference on the 7 point Likert scale, with 80% power at 0.05% significance 45 patients will be needed in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients from 18-75 years
2. A history of symptoms of bladder pain/discomfort described as suprapubic pain related to bladder filling, accompanied by other symptoms such as daytime and/or nighttime frequency in the absence of infection or other pathology, with or without the typical cystoscopic findings of interstitial cystitis
3. Patients willing and able to complete the necessary questionnaires

Exclusion Criteria:

1. Patients with transitional cell carcinoma of the bladder or other significant malignancy
2. Pregnant women
3. Breastfeading women
4. Patients with significant bacteriuria
5. Patients with hematuria
6. Neurogenic bladder
7. Patients with indwelling catheters
8. Chronic bacterial prostatitis
9. Currently receiving or having received investigational drugs thirty (30) days or less prior to screening
10. Currently receiving or having had prior therapy with intravesical treatment (eg. Uracyst, Cystistat®, heparin or BCG)
11. Receiving therapy for less than three months with antidepressants, antihistaminics, hormonal agonists or antagonists; hence patient not stabilized on therapy. (Stable therapy defined as continuous treatment for at least three months.)
12. IC symptoms relieved by antimicrobials, anticholinergics or antispasmodics
13. Functional Bladder capacity of greater than 400 ml
14. Neurologic disease affecting bladder function; any previous surgery or procedure having affected bladder function
15. Current diagnosis of chemical, tuberculous or radiation cystitis
16. bladder or lower ureteral calculi
17. History of cancer within the last five years other than adequately treated non-melanoma skin cancers
18. Active sexual transmitted disease
19. Current vaginitis
20. Endometriosis
21. Any condition/disease which in the opinion of the investigator could interfere with patient compliance and/ or interfere with the interpretation of the treatment results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Global response assessment scale | 4 weeks after last treatment
  Primary endpoint: Global response assessment scale.
  This is a 7 point scale asking: As compared to when you started the current study, how would you rate your overall bladder symptoms now? Seven response options are given to the patient: Markedly worse, moderately worse, slightly worse, no change, slightly improved, moderately improved, markedly improved.

SECONDARY OUTCOMES:
Urinary Frequency | 4 weeks after last treatment
  * Frequency measured as the mean frequency on a 3 day micturition diary
  * Nocturia episodes as the mean number of nocturia episodes on a 3 day micturition diary
  * Functional bladder capacity measured as the mean bladder capacity measured on a 3 day micturition diary
  * VAS pain scale
  * O'Leary -Sant scale
Nocturia Episodes | 4 weeks after last treatment
  Nocturia measured on 3 day micturition diary
Functional bladder capacity | 4 weeks after last treatment
  bladder capacity measured on 3 day micturition diary
VAS pain scale | 4 weeks after last treatment
  visual analogue pain scale
O'Leary Sant | 4 weeks after last treatment
  O'Leary Sant questionnaire score

OTHER OUTCOMES:
Drop-out | any time during study
  patients refusing further treatment because of intolerance to the intravesical treatment of by lack of improvement

CONTACTS AND LOCATIONS:
Overall Officials: Dirk JM De Ridder, MD, PhD, Principal Investigator — University Hospitals KU Leuven
Locations (1):
- Urology, University Hospitals KU Leuven, Leuven, Belgium

REFERENCES:
- [Background] Tutolo M, Ammirati E, Castagna G, Klockaerts K, Plancke H, Ost D, Van der Aa F, De Ridder D. A prospective randomized controlled multicentre trial comparing intravesical DMSO and chondroitin sulphate 2% for painful bladder syndrome/interstitial cystitis. Int Braz J Urol. 2017 Jan-Feb;43(1):134-141. doi: 10.1590/S1677-5538.IBJU.2016.0302. PMID 28124536